CLINICAL TRIAL: NCT01405950
Title: Single-Dose, Phase 1b Study to Assess Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics of Tizanidine at 4 Different Oral Dose Levels in Pediatric Subjects With Mild to Moderate Spasticity Due to Cerebral Palsy
Brief Title: Phase 1b Study of Tizanidine in Pediatric Patients With Cerebral Palsy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Please see 'Further study details as provided by Acorda Therapeutics' for explanation of why study stopped.
Sponsor: Acorda Therapeutics (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT10-ZC-08
Record Dates: First submitted 2011-07-25; First posted 2011-07-29 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Spasticity Due to Cerebral Palsy
MeSH Terms: interventions — tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1 (Experimental)
  Interventions: Drug: Zanaflex Capsules
- Dose Level 2 (Experimental)
  Interventions: Drug: Zanaflex Capsules
- Dose Level 3 (Experimental)
  Interventions: Drug: Zanaflex Capsules
- Dose Level 4 (Experimental)
  Interventions: Drug: Zanaflex Capsules

INTERVENTIONS:
Drug: Zanaflex Capsules — 0.025 mg/kg
  Other Names: tizanidine HCI (hydrochloride)
  Arms: Dose Level 1
Drug: Zanaflex Capsules — 0.05 mg/kg
  Other Names: tizanidine HCI (hydrochloride)
  Arms: Dose Level 2
Drug: Zanaflex Capsules — 0.075 mg/kg
  Other Names: tizanidine HCI (hydrochloride)
  Arms: Dose Level 3
Drug: Zanaflex Capsules — 0.1 mg/kg
  Other Names: tizanidine HCI (hydrochloride)
  Arms: Dose Level 4

SUMMARY:
A Single-Dose, Phase 1b, Multicenter, Open-Label Study to Assess the Pharmacokinetics, Safety and Tolerability, and Pharmacodynamics of Tizanidine at 4 Different Oral Dose Levels in Pediatric Subjects 2 to 16 Years Old With Mild to Moderate Spasticity Due to Cerebral Palsy.

DETAILED DESCRIPTION:
Evaluation of the study's progress after the amendment remained challenging with continued pre-screen failures noted in areas of Botox injection inclusion; family participation refusal / disinterest and gastric or jejunostomy tube placement. A third protocol amendment to improve enrollment was discussed with the Investigators who did not believe further amendment would overcome the barriers expressed by parents that would subject their children to an intense study time commitment without direct benefit. The investigative sites were notified that the study was closed to enrollment March 27, 2012.

ELIGIBILITY:
Inclusion Criteria:

* Have clinically diagnosed spasticity resulting from cerebral palsy
* Have a motor disability resulting from a static, nonprogressive brain injury or malformation occurring prenatally or before the age of 2 years
* Have mild to moderate spasticity at screening
* Have a parent or legally accepted representative able to understand and comply with study requirements who voluntarily provides informed consent and agrees to be primarily responsible for adhering to the requirements of the study

Exclusion Criteria:

* Have a history of hypersensitivity or allergic reaction to tizanidine or any of the capsule components
* Have dietary restrictions or food allergies that conflict with a standardized meal
* Have clinically significant psychiatric, gastrointestinal, pulmonary, hematologic, endocrine, cardiovascular, renal, or hepatic disease that requires pharmacologic intervention
* Have an ongoing seizure disorder that requires medical therapy

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Henney, PharmD, Study Director — Acorda Therapeutics
Locations (1):
- University of Louisville Department of Neurology dba Kentucky Neuroscience Research Health Care Outpatient Center (HCOC), Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Zanaflex Capsules : 0.025 mg/kg
- Dose Level 2: Zanaflex Capsules : 0.05 mg/kg
- Dose Level 3: Zanaflex Capsules : 0.075 mg/kg
- Dose Level 4: Zanaflex Capsules : 0.1 mg/kg
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 8 | 2 | 0 | 0
Completed | 7 | 2 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 8 | 2 | 10
Age, Customized [Number; unit: participants]
  2-3 years | 3 | 0 | 3
  4-5 years | 1 | 0 | 1
  6-12 years | 3 | 2 | 5
  13-16 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter AUC0-8 (Area Under the Concentration-time Curve From Time 0 to 8 Hours) of a Single Dose of Tizanidine at 4 Different Dose Levels in Children and Adolescents With Cerebral Palsy and Mild to Moderate Spasticity.
Description: Baseline: immediately before the standardized meal (i.e., before administration of tizanidine) on dosing day
  0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours after administration of tizanidine
  PK parameters will be derived by using WinNonlin Pro (version 5.0.1 or later, Pharsight Corp).
Time Frame: Baseline and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: Pharmacokinetics Population
Measure: Mean (Standard Error); unit: hour*nanogram/mililiter
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 7 | 2 | 0 | 0
hour*nanogram/mililiter | 5.60 (1.79) | 6.11 (1.29) |  |

2. Secondary Outcome: Pharmacokinetic (PK) Parameter Cmax (Maximum Observed Drug Concentration in Plasma) of a Single Dose of Tizanidine at 4 Different Dose Levels in Children and Adolescents With Cerebral Palsy and Mild to Moderate Spasticity.
Description: as for outcome 1
Time Frame: Baseline and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: Pharmacokinetics Population
Measure: Mean (Standard Error); unit: nanogram/mililiter
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 7 | 2 | 0 | 0
nanogram/mililiter | 1.87 (0.60) | 5.29 (0.05) |  |

ADVERSE EVENTS:
Time Frame: Up to 30 days.
Description: Treatment-emergent adverse events (TEAE) were defined as AEs with date/time of onset (or worsening) on or after the start-date/time of administration of study drug and no more than 1 day after the last dose of study drug.
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/2
Other Adverse Events (participants affected / at risk) | 1/8 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=8) | Dose Level 2 (N=2)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.